CLINICAL TRIAL: NCT06313775
Title: The Feasibility of Local Anesthesia for Bilateral Orchiectomy : a Randomized Controlled Trial
Brief Title: Comparison of Spinal Anesthesia and Spermatic Cord Block for Bilateral Orchiectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sanpasitthiprasong Hospital (Other Government)
Responsible Party: Principal Investigator, Thararat Wanthawong, Principal Investigator of Urology department, Sunpasitthiprasong hospital, Ubonratchathani, Thailand, Sanpasitthiprasong Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPS005
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Orchiectomy; Spermatic Cord Block; Spinal Anesthesia; Pain Score; Prostate Cancer
Keywords: Prostate cancer; CaP; Bilateral orchiectomy; Spermatic cord block; pain score; spinal anesthesia
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Castration

STUDY DESIGN:
Intervention Model Description: Simple random sampling
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia (Active Comparator): spinal anesthesia : 0.5%hyperbaric bupivacaine 10-15 mg/dose injected at L3-L5
  Interventions: Procedure: bilateral orchiectomy
- spermatic cord block (Experimental): 1%Xylocaine with adrenaline (Max 7 mg/kg/dose) divided to inject into each side of the spermatic cord 6-8 ml and infiltration into the scrotal incision area 3-4 ml.
  Interventions: Procedure: bilateral orchiectomy

INTERVENTIONS:
Procedure: bilateral orchiectomy — Bilateral simple orchiectomy is the surgical removal of both testicles through an incision in the scrotum.

SUMMARY:
The goal of this randomized controlled trial is to compare intraoperative pain score, Morphine consumption during 6 and 12 hour after surgery, and postoperative complications between SA and SCB groups in metastatic prostate cancer patient. The main question it aims to answer are:

• Is there a difference in the level of pain during bilateral orchiectomy between spinal anesthesia and spermatic cord block?

Participants will undergo bilateral orchidectomy. They will be randomly assigned to two groups: the group receiving spinal anesthesia and the group receiving spermatic cord block If there is a comparison group: Researchers will compare intraoperative pain score, Morphine consumption during 6 and 12 hour after surgery, and postoperative complications in both groups of patients.

DETAILED DESCRIPTION:
Objective : To compare intraoperative pain score, Morphine consumption during 6 and 12 hour after surgery, and postoperative complications between SA and SCB groups.

Material and Method : This Randomized Controlled Trial that collected data from prostate cancer patients who underwent orchiectomy in our institution. Patients were randomly divided into two groups; SA and SCB. Data was collected on intraoperative pain score, 1 hour post-surgery, Morphine consumption during 6 and 12 hour after surgery and complications. All data was statistically analyzed using Independent t-test and Fisher's exact test.

Inclusion criteria : Patients of all ages diagnosed with prostate cancer undergoing treatment with bilateral orchiectomy.

Exclusion criteria :

1. Patients with a history of Xylocaine allergy.
2. Patients with uncorrected bleeding disorders.
3. Patients with paralysis or neurosensory deficits
4. Patients with dementia or cerebrovascular accidents (strokes) that impair communication.
5. Patients with contraindications for spinal anesthesia, including:

   * Patient refusal of spinal anesthesia.
   * Infection at the site of spinal injection.
   * Allergy to specific types of local anesthetics, such as Hyperbaric bupivacaine.
   * Inability of the patient to cooperate with the spinal anesthetic procedure.
   * Suspicion of high intracranial pressure based on abnormal physical examination.
   * Aortic stenosis with fixed cardiac output.
   * Low platelet count.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages diagnosed with prostate cancer undergoing treatment with bilateral orchiectomy

Exclusion Criteria:

1. Patients with a history of Xylocaine allergy.
2. Patients with uncorrected bleeding disorders.
3. Patients with paralysis or neurosensory deficits
4. Patients with dementia or cerebrovascular accidents (strokes) that impair communication.
5. Patients with contraindications for epidural anesthesia, including:

   * Patient refusal of spinal anesthesia.
   * Infection at the site of spinal injection.
   * Allergy to specific types of local anesthetics, such as Hyperbaric bupivacaine.
   * Inability of the patient to cooperate with the spinal anethetic procedure.
   * Suspicion of high intracranial pressure based on abnormal physical examination.
   * Aortic stenosis with fixed cardiac output.
   * Low platelet count.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
intraoperative pain score | Immediate postoperative assessment
  Pain assessment is done using the verbal numerical rating scale, where patients rate their pain level from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain imaginable, without using any materials or equipment.

SECONDARY OUTCOMES:
post-operative pain score | 1 hour after surgery
  Pain assessment is done using the verbal numerical rating scale, where patients rate their pain level from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain imaginable, without using any materials or equipment.
morphine consumption | during 6 and 12 hour after surgery
  Morphine consumption after surgery
post-operative complications | 24 hour after surgery
  Postoperative complications assessment such as acute urinary retention and neurological complications like radiculopathy, neurological deficits, cauda equina syndrome, and paraplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Thararat Wanthawong, MD, Principal Investigator — Sanpasitthiprasong Hospital; Wattanachai Ungjaroenwathana, MD, Principal Investigator — Sanpasitthiprasong Hospital; Sahachart Atichosakun, MD, Principal Investigator — Sanpasitthiprasong Hospital; Rawisara Hongkrisadakorn, MD, Principal Investigator — Sanpasitthiprasong Hospital
Locations (1):
- Sanpasitthiprasong hospital, Ubon Ratchathani, Thailand

IPD SHARING:
Plan to Share IPD: No